CLINICAL TRIAL: NCT02322931
Title: Intra-operative Use of C-arm Cone-beam CT for Quality Assurance of Low-dose-rate Prostate Brachytherapy Dose Delivery
Brief Title: C-arm Cone-beam CT in Prostate Brachytherapy
Acronym: C-arm
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: British Columbia Cancer Agency (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: H14-02658
Record Dates: First submitted 2014-12-12; First posted 2014-12-23 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Imaging interventions (Experimental): Eligible patients who consent to participate in this study will undergo a combination of 4 different imaging interventions (based on the group they're in, as described in the protocol), intra-operatively, in addition to their standard LDR brachytherapy treatment.
  Interventions: Procedure: Intra-operative C-arm CT imaging

INTERVENTIONS:
Procedure: Intra-operative C-arm CT imaging — 1. Two intra-operative C-arm 3D reconstruction scans with the Ziehm Vision FD Vario 3D immediately after treatment implantation, once with the TRUS probe inserted and once with the TRUS probe removed. This involves approximately 10 fluoroscopy snapshots of the prostate.
  2. Two TRUS Sagittal B-mode sweeps and two TRUS axial B-mode sweeps, once mid-way, i.e. after implanting a sub-set of the seeds, and once at the end of the implantation procedure.
  3. One Cine loop C-arm scan in the sagittal plane while retracting the probe.
  4. One 3D C-arm scan immediately after the treatment, with the TRUS probe removed and the patient in the supine position (i.e. legs down).

SUMMARY:
The investigators will assess the feasibility of intraoperative use of C-arm cone-beam CT imaging for intraoperative dosimetric evaluation in prostate low-dose-rate (LDR) brachytherapy. Patients recruited are those who will receive standard LDR brachytherapy for prostate cancer treatment. Consenting patients will undergo additional 3D C-arm cone-beam CT imaging (3D C-arm) and motorized trans-rectal ultrasound (TRUS). Volumetric and dosimetric measures will be compared to those using the standard Day-0 CT images. The investigators hope that the intraoperative 3D C-arm provides quality assurance measures sufficient to eliminate the need for Day-0 CT LDR brachytherapy and provide the opportunity for intraoperative modification of seed delivery plan.

DETAILED DESCRIPTION:
1. Objectives

   * The primary objective of this study is to determine the feasibility of replacing Day-0 CT with intra-operative 3D C-arm imaging. The main benefit of this change is to receive immediate feedback on the quality of treatment. This can lead to the possibility of performing "live" adjustments to the treatment plan based on feedback of actual seed positions achieved after implantation.
   * Secondly, by replacing Day-0 CT, a separate scan performed in a different site will be eliminated from the treatment procedure, freeing up the CT scanner for other clinical uses
2. Hypotheses

   * Primary hypothesis: Intraoperative use of 3D C-arm cone-beam CT can eliminate the need for Day-0 CT for post-implant dosimetry in prostate LDR brachytherapy by providing similar or improved dosimetric accuracy
   * Secondary hypothesis 1: Dosimetric values obtained with the TRUS probe inside the rectum are not significantly different from those measured when the probe is outside the rectum
   * Secondary hypothesis 2: Sagittal TRUS imaging provides better seed and boudnary detection for dosimetric purposes compared to transverse imaging
3. Justification

   Standard post-implant quality assessment at the BC Cancer Agency involves a pelvic CT 2-3 hours after treatment. This scan is performed outside the operating room, in a different location. As a result, it is not possible to receive immediate feedback on the quality of treatment. Furthermore, soft tissue visualization is poor in CT imaging and contouring variability is large. The use of other imaging modalities such as ultrasound would be beneficial. However, since the scan is performed at a different time, and with the patient in a different position, registering the images would be challenging.

   Intra-operative C-arm CT imaging would provide immediate feedback on the quality of treatment, provide the opportunity of using information from intra-operative ultrasound imaging for soft tissue visualization, and eliminate the need for a separate scan in a different location.
4. Research method

   Patients who are receiving low-dose-rate brachytherapy and consent to participate will undergo the additional imaging interventions described in section 5.7 of the application.

   Patients will also undergo a pelvic CT as the standard of care.

   To limit patient exposure to additional radiation dose, the investigators will divide the participants into 3 groups, each of which will receive a portion of the abovementioned scans. Details are described in the attached protocol.

   Seed locations will be identified on the 3D C-arm volume. The prostate volume on the TRUS images will be delineated and the contours will be mapped onto the 3D C-arm volume to compute standard dosimetric parameters (V100, D90). Seeds and contours will be outlined on the corresponding Day-0 CT and standard dosimetric parameters will be computed. Day-0 CT will be contoured by multiple observers to compute variability in the resulting dosimetric parameters. Dosimetric values from the 3D C-arm will be compared to those of Day-0 CT and their intra-observer variability.

   The seeds will be identified on 3D C-arm volumes with the TRUS probe inserted and retracted to create two seed clouds. Corresponding seeds will be matched. The difference between the seed locations in the two seed clouds will be used to model the prostate deformation due to the presence and absence of the TRUS probe.
5. Statistical analysis This is mainly a descriptive one-arm study. No comparative statistical tests will be applied

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 years of age or older
* Must be able to give informed consent
* Must have been diagnosed with prostate cancer, as determined by a prostate biopsy
* Must not have had any prior history of cancer. Participants that have had some types of skins cancer are still able to participate
* Must be eligible for and receiving low-dose-rate prostate brachytherapy

Exclusion Criteria:

* They are unable to undergo general or spinal anesthesia
* They are on anticoagulation therapy (blood thinners)
* They have had previous radiotherapy to the pelvis

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2015-01; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Dosimetric accuracy | 12 months
  To determine if the intraoperative use of 3D C-arm cone-beam CT can eliminate the need for D-0 Ct for post-implant dosimetry in prostate LDR brachytherapy by providing similar or improved dosimetric accuracy

SECONDARY OUTCOMES:
Dosimetric values | 12 months
  To determine if the dosimetric values obtained with the TRUS probe inside the rectum are significantly different from those measured when the probe is outside the rectum
Seed and boundary detection | 12 months
  To determine if Sagittal TRUS imaging provides better seed and boundary detection for dosimetric purposes compared to transverse imaging

CONTACTS AND LOCATIONS:
Overall Officials: William J Morris, MD, Principal Investigator — British Columbia Cancer Agency
Locations (1):
- British Columbia Cancer Agency, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Blasko JC, Mate T, Sylvester JE, Grimm PD, Cavanagh W. Brachytherapy for carcinoma of the prostate: techniques, patient selection, and clinical outcomes. Semin Radiat Oncol. 2002 Jan;12(1):81-94. doi: 10.1053/srao.2002.28667. PMID 11813153
- [Background] Chng N, Spadinger I, Morris WJ, Usmani N, Salcudean S. Prostate brachytherapy postimplant dosimetry: automatic plan reconstruction of stranded implants. Med Phys. 2011 Jan;38(1):327-42. doi: 10.1118/1.3525839. PMID 21361201
- [Background] Dubois DF, Prestidge BR, Hotchkiss LA, Prete JJ, Bice WS Jr. Intraobserver and interobserver variability of MR imaging- and CT-derived prostate volumes after transperineal interstitial permanent prostate brachytherapy. Radiology. 1998 Jun;207(3):785-9. doi: 10.1148/radiology.207.3.9609905.
- [Background] Mahdavi SS, Chng N, Spadinger I, Morris WJ, Salcudean SE. Semi-automatic segmentation for prostate interventions. Med Image Anal. 2011 Apr;15(2):226-37. doi: 10.1016/j.media.2010.10.002. Epub 2010 Oct 26. PMID 21084216
- [Background] Mahdavi SS, Spadinger I, Chng N, Salcudean SE, Morris WJ. Semiautomatic segmentation for prostate brachytherapy: dosimetric evaluation. Brachytherapy. 2013 Jan-Feb;12(1):65-76. doi: 10.1016/j.brachy.2011.07.007. Epub 2011 Sep 25. PMID 21944824
- [Background] Moradi M, Mahdavi SS, Dehghan E, Lobo JR, Deshmukh S, Morris WJ, Fichtinger G, Salcudean ST. Seed localization in ultrasound and registration to C-arm fluoroscopy using matched needle tracks for prostate brachytherapy. IEEE Trans Biomed Eng. 2012 Sep;59(9):2558-67. doi: 10.1109/TBME.2012.2206808. Epub 2012 Jun 29. PMID 22759435
- [Background] Morris WJ, Keyes M, Spadinger I, Kwan W, Liu M, McKenzie M, Pai H, Pickles T, Tyldesley S. Population-based 10-year oncologic outcomes after low-dose-rate brachytherapy for low-risk and intermediate-risk prostate cancer. Cancer. 2013 Apr 15;119(8):1537-46. doi: 10.1002/cncr.27911. Epub 2012 Dec 26. PMID 23280183
- [Background] Narayana V, Roberson PL, Pu AT, Sandler H, Winfield RH, McLaughlin PW. Impact of differences in ultrasound and computed tomography volumes on treatment planning of permanent prostate implants. Int J Radiat Oncol Biol Phys. 1997 Mar 15;37(5):1181-5. doi: 10.1016/s0360-3016(96)00618-9. PMID 9169829
- [Background] Nath R, Bice WS, Butler WM, Chen Z, Meigooni AS, Narayana V, Rivard MJ, Yu Y; American Association of Physicists in Medicine. AAPM recommendations on dose prescription and reporting methods for permanent interstitial brachytherapy for prostate cancer: report of Task Group 137. Med Phys. 2009 Nov;36(11):5310-22. doi: 10.1118/1.3246613. PMID 19994539
- [Background] Roach M 3rd, Faillace-Akazawa P, Malfatti C, Holland J, Hricak H. Prostate volumes defined by magnetic resonance imaging and computerized tomographic scans for three-dimensional conformal radiotherapy. Int J Radiat Oncol Biol Phys. 1996 Jul 15;35(5):1011-8. doi: 10.1016/0360-3016(96)00232-5. PMID 8751410
- [Background] Smith WL, Lewis C, Bauman G, Rodrigues G, D'Souza D, Ash R, Ho D, Venkatesan V, Downey D, Fenster A. Prostate volume contouring: a 3D analysis of segmentation using 3DTRUS, CT, and MR. Int J Radiat Oncol Biol Phys. 2007 Mar 15;67(4):1238-47. doi: 10.1016/j.ijrobp.2006.11.027. PMID 17336224
- [Background] Bice WS Jr, Prestidge BR, Grimm PD, Friedland JL, Feygelman V, Roach M 3rd, Prete JJ, Dubois DF, Blasko JC. Centralized multiinstitutional postimplant analysis for interstitial prostate brachytherapy. Int J Radiat Oncol Biol Phys. 1998 Jul 1;41(4):921-7. doi: 10.1016/s0360-3016(98)90123-7. PMID 9652858